CLINICAL TRIAL: NCT00595673
Title: Safety and Efficacy Study of PB127 Ultrasound Contrast Agent in Patients With Suspected Coronary Artery Disease 007
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Point Biomedical (Industry)
Responsible Party: Tom Ottoboni/Chief Operating Officer, POINT Biomedical Corp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 127-007
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-07

CONDITIONS: Coronary Artery Disease
Keywords: Perfusion; Echocardiograpy; SPECT; angiography; Chest pain
MeSH Terms: conditions — Coronary Artery Disease; Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: PB127 for injectable suspension — 0.175 mg/kg diluted in 150 mL Dextrose in Water 5% in glass bottles to be infused at 250 mL/hour until stead state achieve, 150 mL/hour during rest image acquisition, and 100-150 mL/hr during stress image acquistion. Single IV infusion, not to exceed 60 minutes.
  Other Names: CARDIOsphere®

SUMMARY:
This trial is to compare PB127 echocardiography to other heart imaging studies.

ELIGIBILITY:
Inclusion Criteria:

Stratum 1:

1. Able to provide written informed consent
2. Low (less than 10%) pre-test probability of CAD (Appendix D)
3. Scheduled for clinically indicated stress echocardiography or stress SPECT within the 14 days prior to or following Study Day 1 (prior to coronary angiography) or coronary angiography within the 7 days following Study Day 1
4. Technically adequate unreconstructed stress SPECT data or scheduled for clinically indicated stress SPECT within 14 days of Study Day 1 and prior to coronary angiography
5. Adequate visualization of all myocardial segments in at least one view during non-contrast echocardiography (See Section 5.3.1)
6. No evidence of a right-to-left shunt during non-contrast echocardiography

Stratum 2:

1. Able to provide written informed consent
2. Intermediate (10% to 90%) pre-test probability of CAD (Appendix D)
3. Scheduled for clinically indicated coronary angiography within the 7 days following Study Day 1
4. Technically adequate unreconstructed stress SPECT data or scheduled for stress SPECT within 14 days of Study Day 1 and prior to coronary angiography
5. Adequate visualization of all myocardial segments in at least one view during non-contrast echocardiography (See Section 5.3.1)
6. No evidence of a right-to-left shunt during non-contrast echocardiography

Stratum 3:

1. Able to provide written informed consent
2. High (greater than 90%) pre-test probability of CAD (Appendix D)
3. Scheduled for clinically indicated coronary angiography within the 7 days following Study Day 1
4. Technically adequate unreconstructed stress SPECT data or scheduled for stress SPECT within 14 days of Study Day 1 and prior to coronary angiography
5. Adequate visualization of all myocardial segments in at least one view during non-contrast echocardiography (See Section 5.3.1)
6. No evidence of a right-to-left shunt during non-contrast echocardiography

Exclusion Criteria:

1. Women who are pregnant or lactating
2. Known hypersensitivity or known contraindication to:

   1. Dipyridamole
   2. Ultrasound contrast agents (including PB127 and excipients)
   3. Blood, blood products, albumin, egg, or protein
3. Use of caffeine or xanthine containing products within the 24 hours prior to PB127 MCE
4. Previous exposure to PB127 Ultrasound Contrast Agent
5. Heart transplant
6. Known right-to-left shunt including atrial septal defect
7. Current or history of uncontrolled ventricular tachycardia
8. Current atrial fibrillation, atrial tachycardia, or atrial flutter
9. Pacemaker or defibrillator
10. Unstable cardiac status

    1. Unstable angina grade CCS Class IV severity with ongoing symptoms and/or ongoing infusion of intravenous nitroglycerin (See Appendix F)
    2. Second-degree or greater heart block
    3. Frequent (>60/hour) or symptomatic ventricular ectopics at baseline
    4. Hypertension (SPB >200 and/or DBP >110 mmHg on two consecutive readings within one hour of PB127 MCE)
    5. Hypotension (SPB <90 mmHg)
    6. Severe aortic stenosis (>100 mmHg peak transvalvar gradient or <0.6 cm2 estimated valve area)
    7. Pulmonary edema within the 7 days prior to Study Day 1
    8. Resting oxygen saturation of less than 90%
    9. Q-wave myocardial infarction within the 7 days prior to Study Day 1
    10. PTCA or CABG within the 7 days prior to Study Day 1
11. Chronic Obstructive Pulmonary Disease (COPD) or bronchospastic airway disease which, in the opinion of the Investigator, is significant enough to contraindicate dipyridamole
12. Known history of severe pulmonary hypertension characterized by estimated pulmonary artery systolic pressure of >50 mmHg
13. Use of intravenous or intracoronary contrast agent other than thallium or technetium within the 24 hours prior to Study Day 1
14. Liver disease (i.e., current or previous hepatic viral infection, chronic hepatitis) characterized by one or more of the following

    1. Current jaundice
    2. Elevated bilirubin > upper limit of normal
    3. Currently elevated hepatic enzymes > 2X upper limit of normal
15. Medical conditions or other circumstances that would significantly decrease the chances of obtaining reliable data or achieving the study objectives (i.e., drug dependence, psychiatric disorder, dementia, or associated illness), extenuating circumstances, medical conditions that make it unlikely that a patient can complete the clinical trial or follow-up evaluations, or other reasons for expected poor compliance with the Investigator's instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2002-07; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
To demonstrate the non-inferiority of the diagnostic performance of PB127 MCE versus stress SPECT in the detection and/or exclusion of significant obstructive CAD as defined by QCA or qualifying clinical outcome. | 90 days

SECONDARY OUTCOMES:
To assess the concordance of PB127 MCE with stress SPECT in differentiating between reversible vs. fixed defects in patients with significant obstructive CAD | 28 days
To compare the diagnostic performance of PB127 MCE with stress SPECT in identifying the location of stenosis as identified by coronary angiography. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ehlgen, MD, PhD, Study Director — POINT Biomedical Corp.
Locations (19):
- United States (19):
  - Heartcare, P.C., Scottsdale, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of California San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Krannert Institute of Cardiology, Indianapolis, Indiana
  - The Center for Cardiovascular Studies Kramer & Crouse Cardiology, Shawnee Mission, Kansas
  - Androscoggin Cardiovascular Associates, Auburn, Maine
  - Maine Cardiology Associates, South Portland, Maine
  - Cardiovascular Consultants, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - St. Luke's Roosevelt Hospital Echocardiography Lab, New York, New York
  - Mount Sinai Hospital, New York, New York
  - MidWest Cardiologist Research, Columbus, Ohio
  - Endovascular Research, LLC, Eugene, Oregon
  - Austin Heart, Austin, Texas
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - Methodist DeBakery Heart Center Cardiovascular Imaging Institute, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Inland Cardiology, Spokane, Washington